CLINICAL TRIAL: NCT05861310
Title: Effectivity and Safety of Metronidazole 1% Cream in Rosacea Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Collaborators: Science and Technology Park, Center of Innovation Technologies for Human Health (Industry)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, SpKK - Head of Cosmetic Dermatology Division, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EffectivityofMetro1%Cre
Record Dates: First submitted 2023-04-06; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Rosacea
Keywords: Rosacea; Erythema
MeSH Terms: conditions — Rosacea; Erythema | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Each research subject will receive a different cream and will be given randomly according to a computer program by a statistician. The control group will receive placebo cream (without the drug substance) and the comparison group will receive metronidazole 1% cream. The cream is used for 2 months and will be evaluated every 28 days.
Who Masked: Outcomes Assessor
Masking Description: The investigator who evaluated the outcomes assessor will be blinded to the treatment allocation until the end of data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole 1% Group (Experimental): Metronidazole 1% cream is applied to the entire face twice a day. Giving cream in the morning and at night. Evaluation will be carried out on days 28 and 56.
  Interventions: Drug: Metronidazole 1% Cream,Top
- Placebo Group (Experimental): Placebo cream (without the drug substance) is applied to the entire face twice a day. Giving cream in the morning and at night. Evaluation will be carried out on days 28 and 56.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole 1% Cream,Top — Cream that has an active ingredient in the form of metronidazole with a content of 1%. At the beginning of the study visit, anamnesis and examination of the skin status were carried out. Skin status includes examination of the degree of erythema with a Clinician Erythema Assessment Scale (CEA) score, examination of skin scrapings for demodex examination, dermoscopy examination, and TEWL (Transepidermal Water Loss) examination. Then the participants were given metronidazole 1% cream which was to be used twice a day in the morning and at night. Evaluation of the therapeutic response will be carried out on days 28 and days 56.
  Other Names: Metronidazole 1%
  Arms: Metronidazole 1% Group
Drug: Placebo — Cream that has not medicine. At the beginning of the study visit, anamnesis and examination of the skin status were carried out. Skin status includes examination of the degree of erythema with a Clinician Erythema Assessment Scale (CEA) score, examination of skin scrapings for demodex examination, dermoscopy examination, and TEWL (Transepidermal Water Loss) examination. Then the research subjects were given Placebo cream (without the drug substance) which was to be used twice a day in the morning and at night. Evaluation of the therapeutic response will be carried out on days 28 and days 56.
  Arms: Placebo Group

SUMMARY:
Rosacea is a chronic inflammatory disease of the central facial region, which can also occur in the neck and chest regions. Microbes that play a role in rosacea are Demodex folliculorum and Helicobactor pylori. On the skin with rosacea have decreased skin barrier function. This clinical study will compare the effectiveness and safety of metronidazole 1% cream as the main therapy in rosacea patients. Participants who will become research subjects are women and men aged 18-60 years who meet the inclusion criteria. Research subjects were divided into 2 groups. The control group will use placebo cream (without the drug substance) and the comparison group will use metronidazole 1% cream.

DETAILED DESCRIPTION:
This study is an experimental study with a double-blind randomized controlled trial (RCT) design for researchers and subjects in male and female patients aged 18-60 years who meet the inclusion criteria. This study used 1% metronidazole cream and placebo cream as a comparison. The creams will then be coded as cream A and cream B. This research will be conducted in two places, namely the Dermatology and Venereology Polyclinic, Division of Cosmetic Dermatology, Cipto Mangunkusumo Hospital (RSCM) and the Dermatology and Venereology Polyclinic, University of Indonesia Hospital (RSUI). The control group will use placebo cream (without the drug substance) and the comparison group will use metronidazole 1% cream. All participants will be evaluated twice on days 28 and days 56. Evaluation of response to therapy that will be assessed includes the degree of erythema with a Clinician Erythema Assessment Scale (CEA) score, examination of skin scrapings for demodex examination, dermoscopy examination, and TEWL (Transepidermal Water Loss) examination.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female, aged 18-60 years
* Diagnosed with rosacea
* The patient agreed to participate in the study and signed a inform consent

Exclusion Criteria:

* Taking corticosteroid therapy (oral or topical)
* Patients with a history of using topical therapy on the face within one month before the study
* Taking metronidazole, clarithromycin, or azithromycin within one month before the study
* Patients who are frequently exposed to ultraviolet (UV) light
* Pregnant or breastfeeding
* Patient and/or family do not agree to participate

Drop Out Criteria:

* Pass away during the clinical trial
* Research subjects were not present when scheduling the action or did not comply with the research protocol.
* Research subjects were not present when scheduling the action or did not comply with the research protocol.
* Suffer from coronavirus disease 2019 (COVID-19) at any time during the trial
* Experience major adverse event(s) caused by topical products or treatments given in the clinical trial (e.g. allergic drug eruption or contact dermatitis). The participants will receive appropriate management if such event occurs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The degree of erythema Examination | Day 0
  The degree of erythema are evaluated with the Clinician Erythema Assessment Scale (CEA) score.
  Based on the score of the Clinician Erythema Assessment Scale (CEA), it has a score of 0 if there is no sign of erythema and a score of 4 if the erythema is moderate-severe.
  The degree of erythema are evaluated with the Clinician Erythema Assessment Scale (CEA) score.
  Based on the score of the Clinician Erythema Assessment Scale (CEA), it has a score of 0 if there is no sign of erythema and a score of 4 if the erythema is moderate-severe.
The degree of erythema Examination | Re-evaluation on days 28
  The degree of erythema are evaluated with the Clinician Erythema Assessment Scale (CEA) score.
  Based on the score of the Clinician Erythema Assessment Scale (CEA), it has a score of 0 if there is no sign of erythema and a score of 4 if the erythema is moderate-severe.
  The degree of erythema are evaluated with the Clinician Erythema Assessment Scale (CEA) score.
  Based on the score of the Clinician Erythema Assessment Scale (CEA), it has a score of 0 if there is no sign of erythema and a score of 4 if the erythema is moderate-severe.
The degree of erythema Examination | Re-evaluation on days 56 post-intervention
  The degree of erythema are evaluated with the Clinician Erythema Assessment Scale (CEA) score.
  Based on the score of the Clinician Erythema Assessment Scale (CEA), it has a score of 0 if there is no sign of erythema and a score of 4 if the erythema is moderate-severe.
  The degree of erythema are evaluated with the Clinician Erythema Assessment Scale (CEA) score.
  Based on the score of the Clinician Erythema Assessment Scale (CEA), it has a score of 0 if there is no sign of erythema and a score of 4 if the erythema is moderate-severe.
Dermoscopy Examination | Day 0
  Skin surface is evaluated by dermoscopy examination. This examination is to see whether there are open comedones surrounded by a thin ring of hyperpigmentation as a picture of Dermodex.
Dermoscopy Examination | Re-evaluation on days 28
  Skin surface is evaluated by dermoscopy examination. This examination is to see whether there are open comedones surrounded by a thin ring of hyperpigmentation as a picture of Dermodex.
Dermoscopy Examination | Re-evaluation on days 56 post-intervention
  Skin surface is evaluated by dermoscopy examination. This examination is to see whether there are open comedones surrounded by a thin ring of hyperpigmentation as a picture of Dermodex.
Demodex Examination | Day 0
  Examination of the amount of demodex on the skin is evaluated by examining skin scrapings.
  In the diagnosis of rosacea, the number of demodex found is more than 5 mites/cm2.
Demodex Examination | Re-evaluation on days 28
  Examination of the amount of demodex on the skin is evaluated by examining skin scrapings.
  In the diagnosis of rosacea, the number of demodex found is more than 5 mites/cm2.
Demodex Examination | Re-evaluation on days 56 post-intervention
  Examination of the amount of demodex on the skin is evaluated by examining skin scrapings.
  In the diagnosis of rosacea, the number of demodex found is more than 5 mites/cm2.
Transepidermal water loss Examination | Day 0, Re-evaluation on days 28 and days 56 post-intervention
  Transepidermal water loss evaluated by the TewameterⓇ. Water evaporation rate in a given area of skin, reported in gram/m²/hour.

CONTACTS AND LOCATIONS:
Overall Officials: Irma Bernadette Sitohang, MD, Principal Investigator — Faculty of Medicine, University of Indonesia; Rinadewi Astriningrum, MD, Principal Investigator — Faculty of Medicine, University of Indonesia; Ika Anggraini, MD, Principal Investigator — Indonesia University of Hospital; Wresti Indriatmi, MD, Principal Investigator — Faculty of Medicine, University of Indonesia; Sutriyo M.Si, Dr, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (2):
- Indonesia (2):
  - Rumah Sakit Umum Pusat Cipto Mangunkusumo, Jakarta, DKI Jakarta
  - Universitas Indonesia of Hospital, Depok, West Java